CLINICAL TRIAL: NCT03722069
Title: A Normal Sodium Diet Preserves Serum Sodium Levels During Treatment of Acute Decompensated Heart Failure
Brief Title: Dietary Sodium Intake in Acute Heart Failure
Acronym: SODIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Fundação de Apoio ao Ensino, Pesquisa e Assistência do Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (Other)
Responsible Party: Principal Investigator, Camila Godoy Fabricio, Master, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2383/2014
Record Dates: First submitted 2018-10-24; First posted 2018-10-26 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure; With Decompensation; Heart Failure，Congestive
Keywords: Hyponatremia; Sodium Intake; Blood Pressure; Sodium Chloride
MeSH Terms: conditions — Heart Failure; Hyponatremia | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low sodium diet (Other): 22 patients were randomized to receive 3 g/day of dietary sodium chloride and a limit of fluid intake of 1000 ml/day.
  Interventions: Other: Low sodium diet
- Normal sodium diet (Other): 22 patients were randomized to receive 7 g/day of dietary sodium chloride and a limit of fluid intake of 1000 ml/day.
  Interventions: Other: Normal sodium diet

INTERVENTIONS:
Other: Low sodium diet — Patients received low sodium diet (3g of sodium chloride/day) and a limit of fluid intake of 1000 ml/day.
  Arms: Low sodium diet
Other: Normal sodium diet — Patients received normal sodium diet (7g of sodium chloride/day) and a limit of fluid intake of 1000 ml/day.
  Arms: Normal sodium diet

SUMMARY:
This study is design to assess two levels of dietary sodium intake in the treatment of patients with Acute Decompensated Heart Failure.

DETAILED DESCRIPTION:
This study aim at assessing the effect of two levels of dietary sodium intake during seven days in hospitalized patients with Acute Decompensated Heart Failure. It is a prospective cohort, randomized, with blinded intervention groups: low sodium diet (the patients will receive 3 g/day of dietary sodium intake), and normal sodium diet (patients will receive 7 g/day of dietary sodium intake). Besides that, both groups will be submitted to a fluid intake limited to 1000 ml/day.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Acute Decompensated Heart Failure diagnosis, filling the Framingham diagnostic criteria, hospitalized at campus Hospital das Clínicas of Ribeirão Preto.

Exclusion Criteria:

* Creatinine clearance <30 ml / min / 1.73 m²;
* Acute coronary syndrome;
* Stroke;
* Dementia;
* Severe cognitive impairment;
* Cancer;
* Decompensated diabetes mellitus;
* Severe liver disease;
* Septic shock or with clinical signs of sepsis;
* Chronic renal parenchymal disease prior to the start of the study;
* ADHF secondary to acute renal failure;
* Nutritional disorders or those who are unable to take oral intake because of vomiting, dysphagia or gastroenteritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-07-20 (Actual); Primary Completion 2017-08-20 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Serum sodium level at day 7 | 7 days
  The difference of the absolute value of serum sodium between the groups in the final evaluation.

SECONDARY OUTCOMES:
Occurrence of hyponatremia | on day 7
  The detection of serum level of sodium bellow 135 mmol/L
Change in body weight | 7 days
  The difference of the absolute value of body weight between the initial and final values.
Change in serum levels of NT-proBNP | 7 days
  The difference of the absolute value of NT-proBNP between the initial and final values, and between groups.
Change in systolic, diastolic and mean blood pressure | 7 days
  The difference of the absolute value of blood pressure between the initial and final values.
Change in heart rate | 7 days
  The difference of the absolute value of heart rate between the initial and final values.
Change in serum levels of creatinine | 7 days
  The difference of the absolute value of creatinine between the initial and final values.
Proportion of patients exhibiting worsening renal function (defined as increased serum creatinine> 0,3 mg / dL) | 7 days
Change in dyspnea sense | 7 days
  Using a visual anologic scale, with values between 0 and 10, where the minimum 0 is the greatest lack of air (worse) and the maximum 10 is the complete breath (better)
Change in well-being sense | 7 days
  Using a visual anologic scale, with values between 0 and 10, where the minimum 0 is the worse you ever felt (worse) and the maximum 10 is feel better than already (better)
Diuretic dosage and other drugs to ADHF during intervention period | 7 days
  What drugs will be used and the quantities.
Rate of hospital readmission | 30 days
Rate of mortality after discharge | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Marcus V Simões, PhD, Principal Investigator — Medical School of Ribeirao Preto, University of Sao Paulo
Locations (1):
- Hospital das Clínicas de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aliti GB, Rabelo ER, Clausell N, Rohde LE, Biolo A, Beck-da-Silva L. Aggressive fluid and sodium restriction in acute decompensated heart failure: a randomized clinical trial. JAMA Intern Med. 2013 Jun 24;173(12):1058-64. doi: 10.1001/jamainternmed.2013.552. PMID 23689381
- [Background] Paterna S, Gaspare P, Fasullo S, Sarullo FM, Di Pasquale P. Normal-sodium diet compared with low-sodium diet in compensated congestive heart failure: is sodium an old enemy or a new friend? Clin Sci (Lond). 2008 Feb;114(3):221-30. doi: 10.1042/CS20070193. PMID 17688420
- [Background] Paterna S, Parrinello G, Cannizzaro S, Fasullo S, Torres D, Sarullo FM, Di Pasquale P. Medium term effects of different dosage of diuretic, sodium, and fluid administration on neurohormonal and clinical outcome in patients with recently compensated heart failure. Am J Cardiol. 2009 Jan 1;103(1):93-102. doi: 10.1016/j.amjcard.2008.08.043. Epub 2008 Oct 17. PMID 19101237
- [Derived] Fabricio CG, Tanaka DM, Souza Gentil JR, Ferreira Amato CA, Marques F, Schwartzmann PV, Schmidt A, Simoes MV. A normal sodium diet preserves serum sodium levels during treatment of acute decompensated heart failure: A prospective, blind and randomized trial. Clin Nutr ESPEN. 2019 Aug;32:145-152. doi: 10.1016/j.clnesp.2019.03.009. Epub 2019 Apr 16. PMID 31221280